CLINICAL TRIAL: NCT03557229
Title: Randomized Controlled Clinical Trial of Antioxidant Therapy in Critically Ill Patients With Septic Shock: Analysis Before and After Treatment of the Oxidative Stress
Brief Title: Clinical Trial of Antioxidant Therapy in Patients With Septic Shock
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American British Cowdray Medical Center (Other)
Responsible Party: Principal Investigator, Alfredo Aisa Alvarez, Principal Investigator, American British Cowdray Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABC-18-19
Record Dates: First submitted 2018-05-11; First posted 2018-06-14 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Oxidative Stress; Septic Shock
Keywords: Oxidative Stress; Sepsis; Treatment; Antioxidant therapy
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Melatonin; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Melatonin (Experimental)
  Interventions: Drug: Melatonin 5 mg
- Vitamin C (Experimental)
  Interventions: Drug: Vitamin C 1 GM Oral Tablet
- Vitamin E (Experimental)
  Interventions: Drug: Vitamin E 400 UNT
- N-acetylcysteine (Experimental)
  Interventions: Drug: N-acetylcysteine
- Control (No Intervention)

INTERVENTIONS:
Drug: Melatonin 5 mg — Oral: 50 mg once daily for 5 days
  Arms: Melatonin
Drug: Vitamin C 1 GM Oral Tablet — Oral: 1 GM every 6 hours for 5 days
  Arms: Vitamin C
Drug: Vitamin E 400 UNT — Oral: 400 UNT every 8 hours for 5 days
  Arms: Vitamin E
Drug: N-acetylcysteine — Oral: 1200 mg every 12 hours for 5 days
  Arms: N-acetylcysteine

SUMMARY:
Sepsis and septic shock are public health problems worldwide that represents an excessive cost for health systems. Despite the great technological and research advances, mortality can reach up to 80% in patients with multiple organ failure (FOM). Therapeutic studies focused on evaluating the usefulness of the use of antioxidants have shown different outcomes and results. This randomized clinical trial in patients with septic shock at two general intensive care units try to evaluate the usefulness of four different antioxidant therapies added to the conventional treatment, which includes: n-acetyl cysteine, vitamin C, vitamin E and melatonin. Measurement of parameters before and after treatment of oxidative stress includes nitrates and nitrites, lipid peroxidation, glutathione peroxidase, glutathione s transferase, extracellular activity of SOD, GSH concentration and evaluation of total antioxidant capacity. The investigators will also evaluate the clinical impact of antioxidant therapy with the SOFA score.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of septic shock in the last 24 hours characterized by refractory hypotension and vasopressor requirement despite sufficient fluid resuscitation (20 mL/kg of colloids or 40 mL/kg of crystalloids) to maintain a blood pressure ≥ 65 mmHg with a lactate> 2 mmol/L.
* Admitted to the ICU of the ABC Medical Center.
* Give informed consent.

Exclusion Criteria:

* Patients who refuse to be included.
* Chronic or recent use of steroids.
* Use of statins.
* Patients receiving some type of antioxidant treatment.
* Any contraindication to the use of vitamin C, vitamin E, n-acetylcysteine or melatonin.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2018-07-23 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Organic failure measurement by the Sequential Organ Failure Assessment Score (SOFA) | Up to 7 days (1 week). From date of randomization and every 24 hours until discharge from the intensive care unit or date of death from any cause, whichever came first, assessed up to 7 days.
  The SOFA score is used to track a person's status during the stay in an intensive care unit (ICU) to determine the extent of a person's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure). The worst physiological variables is collected serially every 24 hours of a patient's ICU admission. The "worst" measurement is defined as the measure that correlated to the highest number of points. The SOFA score ranges from 0 to 24. The investigators are going to evaluate the daily total score and the trend before and after the administration of the therapy.

SECONDARY OUTCOMES:
Nitrates and nitrites levels | Immediately before treatment and 48 hours after therapy
  Oxidative stress
Malondialdehyde levels | Immediately before treatment and 48 hours after therapy
  Lipid peroxidation
Total antioxidant capacity | Immediately before treatment and 48 hours after therapy
  Antioxidant status
Glutathione Peroxidase Enzyme Activity | Immediately before treatment and 48 hours after therapy
  Antioxidant status
Glutathione S-transferase Activity | Immediately before treatment and 48 hours after therapy
  Antioxidant status
Extracellular Superoxide Dismutase Activity | Immediately before treatment and 48 hours after therapy
  Antioxidant status
Glutathione concentration | Immediately before treatment and 48 hours after therapy
  Antioxidant status
Selenium | Immediately before treatment and 48 hours after therapy
  Antioxidant status
Vitamin C | Immediately before treatment and 48 hours after therapy
  Antioxidant status
Thioredoxin | Immediately before treatment and 48 hours after therapy
  Antioxidant status
Carbonylation | Immediately before treatment and 48 hours after therapy
  Pro-oxidant status

OTHER OUTCOMES:
TNF-α | Immediately before treatment and 48 hours after therapy
  Inflammatory Response Pathway
IL-1 | Immediately before treatment and 48 hours after therapy
  Inflammatory Response Pathway
IL-6 | Immediately before treatment and 48 hours after therapy
  Inflammatory Response Pathway
Ionized Ca2+ | Immediately before treatment and 48 hours after therapy
  Electrolytes
Ionized Mg2+ | Immediately before treatment and 48 hours after therapy
  Electrolytes

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Aisa Alvarez, MD, Principal Investigator — American British Cowdray Medical Center
Locations (1):
- Centro Médico ABC, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aisa-Alvarez A, Perez-Torres I, Guarner-Lans V, Manzano-Pech L, Cruz-Soto R, Marquez-Velasco R, Casarez-Alvarado S, Franco-Granillo J, Nunez-Martinez ME, Soto ME. Randomized Clinical Trial of Antioxidant Therapy Patients with Septic Shock and Organ Dysfunction in the ICU: SOFA Score Reduction by Improvement of the Enzymatic and Non-Enzymatic Antioxidant System. Cells. 2023 May 6;12(9):1330. doi: 10.3390/cells12091330. PMID 37174730